CLINICAL TRIAL: NCT03776136
Title: A Multicenter, Open-label, Phase 2 Trial to Assess the Efficacy and Safety of Lenvatinib (E7080/MK-7902) in Combination With Pembrolizumab (MK-3475) in Participants With Advanced Melanoma Previously Exposed to an Anti-PD-1/L1 Agent (LEAP-004)
Brief Title: Efficacy and Safety of Lenvatinib (E7080/MK-7902) Plus Pembrolizumab (MK-3475) for Advanced Melanoma in Anti-Programmed Death-1/Programmed Death-Ligand 1 (PD-1/L1)-Exposed Participants (MK-7902-004/E7080-G000-225/LEAP-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7902-004; MK-7902-004 (Other: MSD Protocol Number); E7080-G000-225 (Other: Eisai Protocol Number); LEAP-004 (Other Grant/Funding Number: MSD); 2018-002518-10 (EudraCT Number)
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Advanced Melanoma
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); programmed cell death ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- lenvatinib plus pembrolizumab (Experimental): Participants receive lenvatinib 20 mg orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W). Pembrolizumab will be administered for up to 35 cycles (approximately 24 months). Lenvatinib will be administered until progressive disease or unacceptable toxicity.
  Interventions: Drug: lenvatinib; Biological: pembrolizumab

INTERVENTIONS:
Drug: lenvatinib — Administered orally once a day during each 21-day cycle.
  Other Names: MK-7902; E7080; LENVIMA™
Biological: pembrolizumab — Administered as an IV infusion on Day 1 Q3W.
  Other Names: MK-3475; Keytruda®

SUMMARY:
This study will evaluate the safety and efficacy of combination therapy of lenvatinib (E7080/MK-7902) and pembrolizumab following approximately 2 years of pembrolizumab therapy and approximately 2 years or more lenvatinib therapy in adult participants with unresectable or advanced melanoma who have been exposed to anti-programmed cell death ligand 1 (PD-1/L1) agents approved for unresectable or metastatic melanoma. No statistical hypothesis will be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed melanoma
* Has unresectable Stage III or Stage IV melanoma per American Joint Committee on Cancer (AJCC) staging system version 8 that is not amenable to local therapy
* Has the presence of ≥1 measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1 as confirmed by BICR.
* Has progressed on treatment with an anti-PD-1/L1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies
* Has submitted pre-trial imaging
* Has an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Has provided a baseline tumor biopsy
* Has resolution of toxic effect(s) of the most recent prior therapy to Grade 1 or less (except alopecia). If participant received major surgery or radiation therapy of >30 Gray (Gy), they must have recovered from the toxicity and/or complications from the Intervention
* Male participants must agree to use approved contraception during the treatment period and for at least 120 days after the last dose of study intervention and refrain from donating sperm during this period
* Female participants are not pregnant and not breastfeeding, and are not a woman of childbearing potential (WOCBP) or are a WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 120 days after the last dose of study intervention
* Has adequate organ function

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment
* Has a known additional malignancy that is progressing or requires active treatment
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has ocular melanoma
* Has known hypersensitivity to active substances or any of their excipients including previous clinically significant hypersensitivity reaction to treatment with another monoclonal antibody
* Has an active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs)
* Has an active infection requiring systemic therapy
* Has known history of Human Immunodeficiency Virus (HIV) or HIV 1/2 antibodies
* Has known history of or is positive for hepatitis B (hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (HCV RNA qualitative] is detected)
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease
* Has a history of active tuberculosis (Bacillus tuberculosis)
* Has presence of a gastrointestinal condition including malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib
* Has had major surgery within 4 weeks prior to first dose of study interventions (adequate wound healing after major surgery must be assessed clinically, independent of time elapsed for eligibility)
* Has a pre-existing Grade ≥3 gastrointestinal or non-gastrointestinal fistula
* Has radiographic evidence of major blood vessel invasion/infiltration
* Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug
* Has clinically significant cardiovascular disease within 12 months from first dose of study drug, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability
* Has received prior radiotherapy within 2 weeks of Cycle 1 Day 1 with the exception of palliative radiotherapy to bone lesions, which is allowed if completed 2 weeks prior to Cycle 1 Day 1
* Has received a live vaccine within 30 days before the first dose of study treatment
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has a history or has current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has had an allogeneic tissue/solid organ transplant
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (23):
- United States (6):
  - Ironwood Cancer & Research Centers ( Site 0312), Chandler, Arizona
  - John Wayne Cancer Institute ( Site 0301), Santa Monica, California
  - Advocate Medical Group-Park Ridge ( Site 0313), Park Ridge, Illinois
  - Southeast Nebraska Cancer Center ( Site 0316), Lincoln, Nebraska
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center ( Site 0317), Dallas, Texas
  - Inova Schar Cancer Institute ( Site 0314), Fairfax, Virginia
- Australia (5):
  - Melanoma Institute Australia ( Site 0152), Wollstonecraft, New South Wales
  - Princess Alexandra Hospital ( Site 0154), Woolloongabba, Queensland
  - Box Hill Hospital ( Site 0157), Box Hill, Victoria
  - Fiona Stanley Hospital ( Site 0156), Perth, Western Australia
  - Lismore Base Hospital ( Site 0153), Lismore
- Canada (4):
  - Sunnybrook Research Institute ( Site 0654), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0655), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0652), Montreal, Quebec
  - McGill University Health Centre ( Site 0651), Montreal, Quebec
- Spain (4):
  - Hospital Clinic i Provincial Barcelona ( Site 0001), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 0003), Madrid
  - Hospital Universitario Virgen de la Macarena ( Site 0004), Seville
  - Hospital General Universitario de Valencia ( Site 0002), Valencia
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset ( Site 0052), Gothenburg
  - Skanes Universitetssjukhus ( Site 0053), Lund
  - Karolinska Universitetssjukhuset ( Site 0051), Solna
  - Norrlands Universitetssjukhus ( Site 0056), Umeå

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Arance A, de la Cruz-Merino L, Petrella TM, Jamal R, Ny L, Carneiro A, Berrocal A, Marquez-Rodas I, Spreafico A, Atkinson V, Costa Svedman F, Mant A, Khattak MA, Mihalcioiu C, Jang S, Cowey CL, Smith AD, Hawk N, Chen K, Diede SJ, Krepler C, Long GV. Phase II LEAP-004 Study of Lenvatinib Plus Pembrolizumab for Melanoma With Confirmed Progression on a Programmed Cell Death Protein-1 or Programmed Death Ligand 1 Inhibitor Given as Monotherapy or in Combination. J Clin Oncol. 2023 Jan 1;41(1):75-85. doi: 10.1200/JCO.22.00221. Epub 2022 Jul 22. PMID 35867951
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenvatinib + Pembrolizumab: Participants received lenvatinib 20 mg orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W). Pembrolizumab was administered for up to 35 cycles (approximately 24 months). Lenvatinib was administered until progressive disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | Lenvatinib + Pembrolizumab
Started | 103
Treated | 103
Completed | 0
Not Completed | 103
Not completed — Death | 85
Not completed — Withdrawal by Subject | 3
Not completed — Sponsor Decision | 15

BASELINE CHARACTERISTICS:
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 98
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants in the analysis population who have a confirmed Complete Response (CR: disappearance of all lesions) or a Partial Response (PR: ≥30% decrease in the sum of target lesion diameters without progression in other lesions) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR). Per protocol, RECIST 1.1 was modified to allow up to 10 target lesions total (up to 5 per organ).
Time Frame: Up to approximately 55 months
Population: All participants who received at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 103
Percentage of Participants | 21.4 [13.9 to 30.5]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from first day of study intervention to the first documented progressive disease (PD) per RECIST 1.1 by BICR, or death from any cause, whichever occurred first. Per protocol, RECIST 1.1 was modified to allow up to 10 target lesions total (up to 5 per organ). PFS was calculated using the nonparametric Kaplan-Meier method; participants who did not experience a PFS event were censored at the last disease assessment, or the last assessment before new anticancer treatment if new treatment was initiated.
Time Frame: Up to approximately 55 months
Population: All participants who received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 103
Months | 4.2 [3.5 to 6.3]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first day of study intervention to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS was calculated using the nonparametric Kaplan-Meier method.
Time Frame: Up to approximately 55 months
Population: All participants who received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 103
Months | 14.0 [10.8 to 18.3]

4. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed Complete Response (CR: disappearance of all lesions) or Partial Response (PR: ≥30% decrease in the sum of target lesion diameters without progression in other lesions) per RECIST 1.1, DOR was defined as the time from first documented CR or PR until progressive disease (PD) or death from any cause, whichever occurs first. Per protocol, RECIST 1.1 was modified to allow up to 10 target lesions total (up to 5 per organ). DOR was calculated using the nonparametric Kaplan-Meier method for censored data.
Time Frame: Up to approximately 55 months
Population: All participants who received at least one dose of study intervention, and who experience a confirmed CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 22
Months | 8.5 [3.2 to 40.8]

5. Secondary Outcome: Area Under the Concentration Time Curve of Lenvatinib From Time 0 to Infinity (AUC 0-inf)
Description: AUC0-inf was defined as the area under the concentration-time curve from time zero extrapolated to infinity. Plasma blood samples collected at specified timepoints, were used to estimate AUC0-inf following Lenvatinib and Pembrolizumab administration. Based on the lenvatinib plasma concentration data obtained on Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1, a protocol specified population PK analysis was performed to characterize the steady state AUC0-inf of lenvatinib when co-administered with pembrolizumab.
Time Frame: Cycle 1 Day 1: 0.5 to 4 hours and 6 to 10 hours postdose; Cycle 1 Day 15: Predose and 2 to 12 hours postdose; Cycle 2 Day 1: Predose, 0.5 to 4 hours, and 6 to 10 hours post-dose (each cycle =21 days)
Population: All participants who received at least one dose of study intervention, and had data available for AUC0-inf.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 103
ng*hr/mL | 3005 (39.5)

6. Secondary Outcome: Number of Participants Who Experience At Least One Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 55 months
Population: All participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 103
Participants | 102

7. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 48 months
Population: All participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 103
Participants | 15

ADVERSE EVENTS:
Time Frame: Up to approximately 55 months
Description: All-cause mortality and adverse events (AE): all participants who received ≥1 dose of treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Lenvatinib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 86/103
Serious Adverse Events (participants affected / at risk) | 48/103
Other Adverse Events (participants affected / at risk) | 101/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=103)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Enteritis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (2)
Proctitis (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (2)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Pelvic abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Horner's syndrome (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (3)
Renal impairment (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=103)
Anaemia (Blood and lymphatic system disorders) | 14 (15)
Neutropenia (Blood and lymphatic system disorders) | 7 (9)
Hypothyroidism (Endocrine disorders) | 37 (39)
Abdominal pain (Gastrointestinal disorders) | 19 (27)
Abdominal pain upper (Gastrointestinal disorders) | 9 (13)
Constipation (Gastrointestinal disorders) | 32 (39)
Diarrhoea (Gastrointestinal disorders) | 50 (123)
Dry mouth (Gastrointestinal disorders) | 15 (18)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (13)
Nausea (Gastrointestinal disorders) | 46 (64)
Stomatitis (Gastrointestinal disorders) | 14 (15)
Toothache (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 28 (51)
Asthenia (General disorders) | 31 (59)
Fatigue (General disorders) | 36 (44)
Mucosal inflammation (General disorders) | 18 (30)
Oedema peripheral (General disorders) | 6 (6)
Pyrexia (General disorders) | 20 (23)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 15 (17)
Alanine aminotransferase increased (Investigations) | 16 (19)
Amylase increased (Investigations) | 10 (15)
Aspartate aminotransferase increased (Investigations) | 13 (18)
Blood alkaline phosphatase increased (Investigations) | 7 (9)
Blood magnesium decreased (Investigations) | 6 (18)
Blood thyroid stimulating hormone increased (Investigations) | 9 (12)
Haemoglobin decreased (Investigations) | 7 (10)
Lipase increased (Investigations) | 14 (14)
Neutrophil count decreased (Investigations) | 6 (6)
Weight decreased (Investigations) | 23 (25)
Decreased appetite (Metabolism and nutrition disorders) | 42 (58)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (15)
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 (23)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (39)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (24)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (12)
Dizziness (Nervous system disorders) | 18 (22)
Dysgeusia (Nervous system disorders) | 12 (15)
Headache (Nervous system disorders) | 29 (56)
Insomnia (Psychiatric disorders) | 11 (12)
Proteinuria (Renal and urinary disorders) | 23 (34)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 22 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (11)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (19)
Rash (Skin and subcutaneous tissue disorders) | 12 (15)
Vitiligo (Skin and subcutaneous tissue disorders) | 6 (6)
Hypertension (Vascular disorders) | 58 (88)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03776136/Prot_SAP_000.pdf